CLINICAL TRIAL: NCT06060171
Title: Pathological Changes in the Cardiovascular System in Valvular Heart Disease: Validation of Non-invasive Markers
Brief Title: Pathological Changes in the Cardiovascular System in Valvular Heart Disease
Acronym: PATH-VHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: British Heart Foundation (Other); Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: 134018
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Septal myocardial biopsies Blood biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Natural history: Natural history of the three common valvular lesions; aortic stenosis, aortic regurgitation and mitral regurgitation. Patients with mild, moderate and severe valvular heart disease (VHD) will be followed up at 1-year to measure progression in remodelling (hypertrophy, ischaemic, scar).
- Multisystem impact of VHD: Patients with severe symptomatic VHD will undergo non-invasive brain and cardiac magnetic resonance imaging (MRI) plus other non-invasive imaging tests to quantify small blood vessels across the cardiovascular system at baseline and at 6 months after surgical aortic valve replacement at which point a myocardial biopsy is taken.
  Interventions: Procedure: Aortic valve intervention
- Response to intervention.: Patients with severe symptomatic VHD undergoing intervention will be followed up at 6 months to assess reverse remodelling after valve intervention. In those undergoing open-heart surgery, a myocardial biopsy will be taken to validate and complement non-invasive imaging.
  Interventions: Procedure: Aortic valve intervention

INTERVENTIONS:
Procedure: Aortic valve intervention — Surgical or transcatheter aortic valve intervention
  Groups: Multisystem impact of VHD; Response to intervention.

SUMMARY:
An observational cohort study of patients recruited presenting with valvular heart disease. The specialized investigations will focus on myocardial remodelling and scar formation/regression and extracardiac micro- and macro-vascular sequelae of valvular heart disease (VHD). The aim is to investigate the natural history of VHD and its ensuing cardiac and extracardiac end organ effects, the impact of existing interventions and the long-term outcome. We hope to establish the underlying causative aetiology of known associated conditions (e.g. vascular dementia) and to determine if extracardiac changes may serve as early biomarkers of prognosis in VHD. Participants will attend for two visits at Barts Heart Centre or Chenies Mews Imaging Centre and will undergo a panel of tests including cross-sectional cardiac imaging, point-of-care microvascular assessment and blood tests. Patient outcome will be assessed by data linkage to hospital episode statistic (HES) data and ONS data (via NHS spine). We aim to identify determinants that will help to improve patient selection and timing of valve intervention based on advanced clinical, blood and/or imaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to provide written informed consent
* Mild, moderate or severe valvular heart disease (Natural history cohort), or severe valvular heart disease planned for surgical/transcatheter intervention (Intervention/Heart-Brain axis cohort).

Exclusion Criteria:

* Participants unwilling to consent.
* Needle phobic patients that would preclude blood taking
* Diagnosis of dilated or hypertrophic cardiomyopathy
* Pregnancy/breast feeding
* Inability to complete the protocol, other conditions that would prevent participation in the study.
* In severe VHD, no more than moderate valve disease other than primary lesion (AS / MR / AR)

Exclusion for the Heart-Brain-Axis Study:

• Participants that have more than moderate epicardial coronary disease (by CT or invasive coronary angiography) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Natural history cohort: Patients with three common valvular lesions: Aortic stenosis, aortic regurgitation and mitral regurgitation
  Multisystem impact of valvular heart disease: Patients with severe symptomatic valvular heart disease referred for surgery
  Response to intervention: Patients with severe symptomatic valvular heart disease undergoing intervention
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Multisystem study: Correlation between capillary density and stress myocardial blood flow in severe valve disease before intervention (at baseline) | Single timepoint
Multisystem study: Correlation between brain blood flow (arterial spin labelling) and stress myocardial blood flow in severe valve disease before intervention (at baseline) | Single timepoint
Intervention study: Change in stress myocardial blood flow from baseline to 6 months after aortic valve replacement | Baseline and 6 months after surgery
Intervention study: Correlation between functional capacity, measured by cardiopulmonary exercise testing and myocardial blood flow and fibrosis by cardiovascular magnetic resonance and histology at baseline and at 6 months after valve replacement | Baseline and 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No